CLINICAL TRIAL: NCT00705146
Title: Comparison of Two Carpometacarpal Stabilizing Splints for People With Thumb Osteoarthritis
Brief Title: CMC (Carpometacarpal) OA (Osteoarthritis) Thumb Splint Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H07-03133
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, carpometacarpal joint; Thumb splints; AUSCAN-HI 3.1; Grip and pinch strength
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comfort Cool Splint (Active Comparator): Comfort Cool(TM) splint, a prefabricated neoprene splint, fit according to the participant's size (S, M, M+, L). Participants instructed to wear the splint when symptomatic, during manual tasks, and at night if desired. Used for 4 weeks.
  Interventions: Device: Comfort Cool thumb splint by North Coast Medical
- Hybrid Custom-made splint (Active Comparator): The Hybrid splint was based on Pat McKee's custom-made splint design, fabricated from neoprene and 1.6 mm Rolyan Aquaplast Watercolors (Bollingbrook, IL). Participants were instructed to wear the splint when symptomatic, during manual tasks, and at night if desired. Splint was worn for 4 weeks.
  Interventions: Device: Custom made thermoplastic & neoprene splint

INTERVENTIONS:
Device: Comfort Cool thumb splint by North Coast Medical — Comfort Cool(TM) splint, a prefabricated neoprene splint, fit according to the participant's size (S, M, M+, L). Participants instructed to wear the splint when symptomatic, during manual tasks, and at night if desired. Used for 4 weeks. Treating therapists did not provide exercises or joint protection education until the final outcome measurement session at 9 weeks.
  Arms: Comfort Cool Splint
Device: Custom made thermoplastic & neoprene splint — The Hybrid splint was based on Pat McKee's custom-made splint design, fabricated from neoprene and 1.6 mm Rolyan Aquaplast Watercolors (Bollingbrook, IL). Participants were instructed to wear the splint when symptomatic, during manual tasks, and at night if desired. Splint was worn for 4 weeks. Treating therapists did not provide exercises or joint protection education until the final outcome measurement session at 9 weeks.
  Arms: Hybrid Custom-made splint

SUMMARY:
Osteoarthritis (OA) of the thumb carpometacarpal (CMC) joint is a common condition that is seen regularly in outpatient occupational therapy and physiotherapy departments. Prevalence rates of symptomatic thumb OA have been found to be as high as 25%. The conservative treatment of choice consists of splinting. There are many different types of thumb splints available, but no specific guidelines as to which is preferred. There is limited evidence to support the benefits of splinting.

The purpose of this study is to compare the effectiveness of two different thumb splints: the Comfort Cool, a prefabricated neoprene splint and a custom made neoprene and thermoplastic thumb splint. These are two of the most commonly prescribed splints in local occupational therapy departments.

DETAILED DESCRIPTION:
Thumb (CMC) osteoarthritis is treated conservatively with splinting. The objectives of splinting the CMC joint include stabilizing the joint, reducing pain symptoms as well as enhancing performance of everyday activities. There is limited evidence to support the effectiveness of splinting in reducing pain and very little evidence to support the effectiveness of thumb splints to enhance function.

This CMC splint comparison study is a cross-over community based study of the effect of two different types of CMC stabilizing splints on patients with thumb OA. The objectives include measuring clients' OA symptoms and function using the Australian Canadian Osteoarthritis Hand Index (AUSCAN-HI 3.1), grip strength, pinch strength and client's personal splint preference on 4 separate occasions in order to compare the two thumb splints. The two splints differ in material and design. One splint is softer and incorporates more of the hand. The evidence gathered will support the effectiveness of specific splint design. It will also provide best practice guidelines for splint selection in clients with CMC OA.

We are using a one group own control cross-over design where outcome measures will be taken at week 1, week 4, week 5 and week 9. Each client will wear both splints for a 4 week period separated by a 1 week wash out period.

Procedure:

First appointment: At the initial visit the client will be randomly assigned to splint order. The client will complete the AUSCAN-HI 3.1, and a grip and pinch strength measurement. The first CMC stabilizing splint will be fabricated and fitted as per normal splinting treatment for clients with CMC OA. The client will be instructed how to wear and care for their splint. General instructions will include wearing the splint for symptomatic use as well as heavy activities.

Second visit: The second visit will take place 4 weeks after the first unless the client needs to come in earlier for a splint adjustment. At this time the AUSCAN-HI 3.1 will be administered again. Grip and pinch strength will also be re-measured.

Third visit: After a one week wash-out period where the client does not wear any splint, they will attend the OT Outpatient department and complete the AUSCAN-HI 3.1, perform a grip and pinch strength measurement. They will be provided with the second CMC stabilizing splint and instructed in a wearing regime and the care of it.

Fourth visit: This will take place at approximately 9 weeks, 4 weeks after wearing the second splint. The AUSCAN-HI 3.1 will be completed for the last time as well as a grip and pinch strength measurement. The client will also be asked their personal splint preference at this time.

Data will be collected and input into the computer.

Note: The procedures for grip and pinch strength measurement will follow the guidelines set out in the ASHT Clinical Assessment Recommendations.

Data Analysis: Data will be analyzed using ANOVA, to determine if there is a significant difference between the 2 splints for OA pain, function, grip strength and personal preference.

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosis of CMC OA
* 45 years or older
* able to read and write in English

Exclusion Criteria:

• previous thumb surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Backman, Ph.D, Principal Investigator — University of British Columbia; Peter Kirk, Ph.D, Study Director — University of British Columbia
Locations (3):
- Canada (3):
  - Campbell River Hospital, Campbell River, British Columbia
  - Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Victoria Island Hand Clinic, Victoria, British Columbia

REFERENCES:
- [Result] Sillem H, Backman CL, Miller WC, Li LC. Comparison of two carpometacarpal stabilizing splints for individuals with thumb osteoarthritis. J Hand Ther. 2011 Jul-Sep;24(3):216-25; quiz 126; discussion 227-30. doi: 10.1016/j.jht.2010.12.004. Epub 2011 Mar 21. PMID 21420278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 outpatient hand therapy departments on Vancouver Island from April 1, 2008 to April 30, 2009.
Groups:
- Hybrid Splint 4 Weeks, 1 Week Washout, Then Comfort Cool Splin: Hybrid splint for 4 weeks, 1 wk washout, then Comfort Cool splint for 4 weeks
- Comfort Cool Splint 4 Weeks, 1 Week Washout, Then Hybrid Splin: Comfort Cool splint for 4 weeks, 1 wk washout, then Hybrid splint for 4 weeks
Period: Overall Study
Arm/Group | Hybrid Splint 4 Weeks, 1 Week Washout, Then Comfort Cool Splin | Comfort Cool Splint 4 Weeks, 1 Week Washout, Then Hybrid Splin
Started | 32 | 24
Completed | 31 | 23
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Hybrid Then Comfort Cool: Hybrid splint for 4 weeks, 1 wk washout, then Comfort Cool splint for 4 weeks
- Comfort Cool Then Hybrid Splint: Comfort Cool splint for 4 weeks, 1 wk washout, then Hybrid splint for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Hybrid Then Comfort Cool | Comfort Cool Then Hybrid Splint | Total
Number analyzed (Participants) | 32 | 24 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 11 | 32
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.84 (8.48) | 65.67 (8.64) | 64.05 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 22 | 51
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 32 | 24 | 56

OUTCOME MEASURES:

1. Primary Outcome: Hand Function
Description: Hand Function was measured with the Australian Canadian Osteoarthritis Hand Index 3.1 (AUSCAN). The AUSCAN is a self-report tool with 15 questions in 3 subscales: pain, function, joint stiffness, and uses an 11-point (0-10) numerical rating scale. The AUSCAN function subscale has 9 items regarding level of difficulty in performing daily tasks such as opening a jar, turning a doorknob, wringing out a washcloth. Possible scores range from 0 to 90. Mean change scores are reported (baseline compared to 4 weeks splint use). Higher scores indicate worse function.
Time Frame: 4 weeks
Population: Pooled participants from both arms from the phase they wore the hybrid splint, then from the phase they wore the comfort cool splint. Mean change scores are reported.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Hybrid Splint: Use of the hybrid splint for 4 weeks
- Comfort Cool Splint: Use of the comfort cool splint for 4 weeks
Arm/Group | Hybrid Splint | Comfort Cool Splint
Number analyzed (Participants) | 56 | 56
units on a scale | 5.54 [0.80 to 10.28] | 2.69 [-1.73 to 7.11]

2. Secondary Outcome: Pain
Description: AUSCAN 3.1 pain subscale. Possible score range is 0 to 50. Lower scores indicate less pain. Change scores are reported (baseline to 4 weeks splint wear) for each of the two splints.
Time Frame: 4 weeks
Population: Pooled all participants for the phase they wore the hybrid, then comfort cool splints, respectively. Mean change scores are reported
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hybrid Splint | Comfort Cool Splint
Number analyzed (Participants) | 56 | 56
units on a scale | 5.69 [2.66 to 8.71] | 2.05 [-0.53 to 4.63]

ADVERSE EVENTS:
Arm/Group | Hybrid Then Comfort Cool | Comfort Cool Then Hybrid Splint
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/24
Other Adverse Events (participants affected / at risk) | 0/32 | 0/24

LIMITATIONS AND CAVEATS:
The main limitation of this cross-over trial was that the therapists who collected the data were not blinded to the splinting intervention, as they were required to fabricate and fit each splint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No